CLINICAL TRIAL: NCT00069576
Title: A Randomized Clinical Trial of Treatment for Mild Gestational Diabetes Mellitus
Brief Title: Gestational Diabetes Mellitus Trial (GDM)
Acronym: GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD36801 - GDM; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD036801 (NIH); U10HD053118 (NIH); U10HD053097 (NIH); U10HD027860 (NIH); U10HD034136 (NIH)
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Diabetes, Gestational
Keywords: Mild gestational diabetes mellitus; Maternal Fetal Medicine Units Network
MeSH Terms: conditions — Diabetes, Gestational | interventions — Nutrition Assessment; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional counseling & self blood glucose monitoring (Active Comparator): Within one week of enrollment, women in the treatment group receive formal nutritional counseling and will be instructed on the technique of self blood glucose monitoring using a memory-based reflectance meter.
  Interventions: Behavioral: nutritional counseling; Behavioral: self blood glucose monitoring
- No treatment (No Intervention): This group will not receive any specific dietary therapy except for written information concerning general nutritional recommendations for normal pregnancy.

INTERVENTIONS:
Behavioral: nutritional counseling
  Arms: Nutritional counseling & self blood glucose monitoring
Behavioral: self blood glucose monitoring
  Arms: Nutritional counseling & self blood glucose monitoring

SUMMARY:
Gestational diabetes mellitus (GDM) is a type of diabetes (high blood sugar) that occurs in pregnant women. This study will determine whether treating pregnant women who have mild GDM improves the health of their babies. The follow-up study will examine whether factors during the previous pregnancy (such as blood sugar during pregnancy) are associated with the woman and her child's health 4-9 years later.

DETAILED DESCRIPTION:
Gestational diabetes mellitus is defined as glucose intolerance of variable severity with onset or first recognition during pregnancy. The definition applies regardless of insulin use for treatment or the persistence of the condition after pregnancy, and does not exclude the possibility that unrecognized glucose intolerance or overt diabetes may have preceded the pregnancy. Pre-existing diabetes substantially contributes to perinatal morbidity and mortality. The association of milder forms of gestational diabetes with adverse pregnancy outcomes, including morbidities such as macrosomia, birth trauma, and neonatal hypoglycemia, remains questionable. While it is likely that maternal glucose intolerances reflect a continuum of risk for adverse outcomes, it is not known whether there is a benefit to identification and subsequent treatment of mild glucose intolerance during pregnancy. This study will determine whether dietary treatment (and insulin as required) for mild GDM will reduce the frequency of neonatal morbidity associated with mild glucose intolerance.

Participants in this study will receive a 50-gram glucose loading test (GLT) between 24 and 30 weeks' gestation. Those with a positive GLT will receive a subsequent 3-hour oral glucose tolerance test (OGTT). Based upon these test results, women will be assigned to 4 groups. Women with a positive GLT and abnormal OGTT will be randomly assigned to receive either nutritional counseling and diet therapy (Group 1) or no specific treatment (Group 2a). Women with a positive GLT but normal OGTT will be enrolled in Group 2b for observation. Women with a negative GLT will be enrolled in Group 3 and will serve as a control group.

Women in Group 1 will receive formal nutritional counseling and will be instructed on the techniques of self blood glucose monitoring. Patients will take daily blood glucose measurements and will be seen at weekly study visits. The study will evaluate birth outcomes, including stillbirth, neonatal hypoglycemia, neonatal hyperinsulinemia, neonatal hyperbilirubinemia, and birth trauma.

The follow-up study will examine if blood sugar levels and treatments during pregnancy influence the health of the mother and child several years later. The study will also examine whether there is a genetic link to the health of the mother and child. The study visit will include blood pressure, body size measurements, blood draw and saliva collection, and questions related to the mother and child's health and environment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Gestational age at enrollment 24 - 31 weeks

Exclusion Criteria:

* Diabetes diagnosed prior to pregnancy
* Abnormal gestational diabetes (>= 135 mg/dl) testing prior to 24 weeks' gestation
* Gestational diabetes in a previous pregnancy
* History of stillbirth or fetal death
* Pregnancy with more than one fetus
* Known major fetal anomaly
* Current or planned corticosteroid therapy
* Asthma requiring medication
* Current or planned beta adrenergic therapy
* Chronic hypertension requiring medication within 6 months of or during pregnancy
* Chronic medical conditions such as HIV/AIDS, kidney disease, or congenital heart disease
* Hematologic or autoimmune disease such as sickle cell disease, other hemoglobinopathies, lupus, or antiphospholipid syndrome
* Maternal or fetal conditions likely to require preterm delivery, such as pre-eclampsia, preterm labor, or intrauterine growth retardation
* Previous or planned tocolytic therapy to induce labor or increase contraction strength

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7381 (Actual)
Dates: Start 2002-10; Primary Completion 2007-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark B. Landon, MD, Study Chair — Ohio State University; Uma Reddy, MD, MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Elizabeth A Thom, Ph.D., Principal Investigator — George Washington University Biostatistics Center
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University - Hutzel Hospital, Detroit, Michigan
  - Columbia University-St. Luke's Hospital, New York, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas-Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Landon MB, Thom E, Spong CY, Gabbe SG, Leindecker S, Johnson F, Lain K, Miodovnik M, Carpenter M. A planned randomized clinical trial of treatment for mild gestational diabetes mellitus. J Matern Fetal Neonatal Med. 2002 Apr;11(4):226-31. doi: 10.1080/jmf.11.4.226.231. PMID 12375675
- [Background] Landon MB, Mele L, Spong CY, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health, and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. The relationship between maternal glycemia and perinatal outcome. Obstet Gynecol. 2011 Feb;117(2 Pt 1):218-224. doi: 10.1097/AOG.0b013e318203ebe0. PMID 21309194
- [Background] Durnwald CP, Mele L, Spong CY, Ramin SM, Varner MW, Rouse DJ, Sciscione A, Catalano P, Saade G, Sorokin Y, Tolosa JE, Casey B, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Glycemic characteristics and neonatal outcomes of women treated for mild gestational diabetes. Obstet Gynecol. 2011 Apr;117(4):819-827. doi: 10.1097/AOG.0b013e31820fc6cf. PMID 21422852
- [Background] Bahado-Singh RO, Mele L, Landon MB, Ramin SM, Carpenter MW, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-fetal Medicine Units Network. Fetal male gender and the benefits of treatment of mild gestational diabetes mellitus. Am J Obstet Gynecol. 2012 May;206(5):422.e1-5. doi: 10.1016/j.ajog.2012.03.015. Epub 2012 Mar 23. PMID 22542118
- [Background] Stuebe AM, Landon MB, Lai Y, Spong CY, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Sciscione A, Catalano P, Harper M, Saade G, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network, Bethesda, MD. Maternal BMI, glucose tolerance, and adverse pregnancy outcomes. Am J Obstet Gynecol. 2012 Jul;207(1):62.e1-7. doi: 10.1016/j.ajog.2012.04.035. Epub 2012 May 2. PMID 22609018
- [Background] Berggren EK, Mele L, Landon MB, Spong CY, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Perinatal outcomes in Hispanic and non-Hispanic white women with mild gestational diabetes. Obstet Gynecol. 2012 Nov;120(5):1099-104. doi: 10.1097/aog.0b013e31827049a5. PMID 23090528
- [Background] Ma KK, Mele L, Landon MB, Spong CY, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. The obstetric and neonatal implications of a low value on the 50-g glucose screening test. Am J Perinatol. 2013 Oct;30(9):715-22. doi: 10.1055/s-0032-1331027. Epub 2012 Dec 27. PMID 23271384
- [Background] Figueroa D, Landon MB, Mele L, Spong CY, Ramin SM, Casey B, Wapner RJ, Varner MW, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Relationship between 1-hour glucose challenge test results and perinatal outcomes. Obstet Gynecol. 2013 Jun;121(6):1241-1247. doi: 10.1097/AOG.0b013e31829277f5. PMID 23812458
- [Background] Costantine MM, Mele L, Landon MB, Spong CY, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network, Bethesda, Maryland. Customized versus population approach for evaluation of fetal overgrowth. Am J Perinatol. 2013 Aug;30(7):565-72. doi: 10.1055/s-0032-1329188. Epub 2012 Nov 12. PMID 23147078
- [Background] Catalano PM, Mele L, Landon MB, Ramin SM, Reddy UM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Saade G, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Inadequate weight gain in overweight and obese pregnant women: what is the effect on fetal growth? Am J Obstet Gynecol. 2014 Aug;211(2):137.e1-7. doi: 10.1016/j.ajog.2014.02.004. Epub 2014 Feb 11. PMID 24530820
- [Background] Sutton AL, Mele L, Landon MB, Ramin SM, Varner MW, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Grobman WA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Delivery timing and cesarean delivery risk in women with mild gestational diabetes mellitus. Am J Obstet Gynecol. 2014 Sep;211(3):244.e1-7. doi: 10.1016/j.ajog.2014.03.005. Epub 2014 Mar 4. PMID 24607755
- [Background] Casey BM, Mele L, Landon MB, Spong CY, Ramin SM, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Catalano P, Harper M, Saade G, Sorokin Y, Peaceman AM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Does maternal body mass index influence treatment effect in women with mild gestational diabetes? Am J Perinatol. 2015 Jan;32(1):93-100. doi: 10.1055/s-0034-1374815. Epub 2014 May 16. PMID 24839145
- [Background] Stuebe AM, Landon MB, Lai Y, Klebanoff M, Ramin SM, Wapner RJ, Varner MW, Rouse DJ, Sciscione A, Catalano P, Saade G, Sorokin Y, Peaceman AM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network, Bethesda, MD. Is There a Threshold Oral Glucose Tolerance Test Value for Predicting Adverse Pregnancy Outcome? Am J Perinatol. 2015 Jul;32(9):833-8. doi: 10.1055/s-0034-1543949. Epub 2015 Jan 16. PMID 25594222
- [Background] Palatnik A, Mele L, Landon MB, Reddy UM, Ramin SM, Carpenter MW, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Saade GR, Caritis SN, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Timing of treatment initiation for mild gestational diabetes mellitus and perinatal outcomes. Am J Obstet Gynecol. 2015 Oct;213(4):560.e1-8. doi: 10.1016/j.ajog.2015.06.022. Epub 2015 Jun 11. PMID 26071920
- [Background] Rice MM, Landon MB, Varner MW, Casey BM, Reddy UM, Wapner RJ, Rouse DJ, Biggio JR Jr, Thorp JM Jr, Chien EK, Saade G, Peaceman AM, Blackwell SC, VanDorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Pregnancy-Associated Hypertension in Glucose-Intolerant Pregnancy and Subsequent Metabolic Syndrome. Obstet Gynecol. 2016 Apr;127(4):771-779. doi: 10.1097/AOG.0000000000001353. PMID 26959208
- [Background] Harper LM, Mele L, Landon MB, Carpenter MW, Ramin SM, Reddy UM, Casey B, Wapner RJ, Varner MW, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Carpenter-Coustan Compared With National Diabetes Data Group Criteria for Diagnosing Gestational Diabetes. Obstet Gynecol. 2016 May;127(5):893-898. doi: 10.1097/AOG.0000000000001383. PMID 27054932
- [Background] Blackwell SC, Landon MB, Mele L, Reddy UM, Casey BM, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Saade G, Caritis SN, Sorokin Y, Grobman WA; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Relationship Between Excessive Gestational Weight Gain and Neonatal Adiposity in Women With Mild Gestational Diabetes Mellitus. Obstet Gynecol. 2016 Dec;128(6):1325-1332. doi: 10.1097/AOG.0000000000001773. PMID 27824768
- [Background] Varner MW, Rice MM, Landon MB, Casey BM, Reddy UM, Wapner RJ, Rouse DJ, Tita ATN, Thorp JM, Chien EK, Saade GR, Peaceman AM, Blackwell SC, Vandorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Pregnancies After the Diagnosis of Mild Gestational Diabetes Mellitus and Risk of Cardiometabolic Disorders. Obstet Gynecol. 2017 Feb;129(2):273-280. doi: 10.1097/AOG.0000000000001863. PMID 28079773
- [Background] Tita ATN, Lai Y, Landon MB, Ramin SM, Casey B, Wapner RJ, Varner MW, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade GR, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Predictive Characteristics of Elevated 1-Hour Glucose Challenge Test Results for Gestational Diabetes. Am J Perinatol. 2017 Dec;34(14):1464-1469. doi: 10.1055/s-0037-1604243. Epub 2017 Jul 19. PMID 28724164
- [Result] Landon MB, Rice MM, Varner MW, Casey BM, Reddy UM, Wapner RJ, Rouse DJ, Biggio JR Jr, Thorp JM, Chien EK, Saade G, Peaceman AM, Blackwell SC, VanDorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. Mild gestational diabetes mellitus and long-term child health. Diabetes Care. 2015 Mar;38(3):445-52. doi: 10.2337/dc14-2159. Epub 2014 Nov 20. PMID 25414152
- [Result] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Derived] Durnwald C, Mele L, Landon MB, Varner MW, Casey BM, Reddy UM, Wapner RJ, Rouse DJ, Tita ATN, Thorp JM Jr, Chien EK, Saade GR, Peaceman AM, Blackwell SC; Eunice Kennedy Shriver National Institute of Child Health Human Development (NICHD) Maternal Fetal Medicine Units (MFMU) Network. Fibroblast Growth Factor 21 and Metabolic Dysfunction in Women with a Prior Glucose-Intolerant Pregnancy. Am J Perinatol. 2021 Nov;38(13):1380-1385. doi: 10.1055/s-0040-1712966. Epub 2020 Jun 23. PMID 32575141
- [Derived] Rice MM, Landon MB, Varner MW, Casey BM, Reddy UM, Wapner RJ, Rouse DJ, Tita ATN, Thorp JM Jr, Chien EK, Saade G, Peaceman AM, Blackwell SC; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Pregnancy-Associated Hypertension and Offspring Cardiometabolic Health. Obstet Gynecol. 2018 Feb;131(2):313-321. doi: 10.1097/AOG.0000000000002433. PMID 29324603
- See also: NICHD Maternal Fetal Medicine Units Network website — http://www.bsc.gwu.edu/mfmu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19,665 pregnant women between 24 weeks 0 days and 30 weeks 6 days gestation with glucose levels greater than or equal to 135mg/dl and less than 200 mg/dl after a 1-hour 50-g glucose loading test were assessed for eligibility in the trial. 500 of the eligible patients consented for teh follow-up study.
Pre-assignment Details: Of the women screened, 7,381 consented to participate but 83 did not complete an oral glucose tolerance test. Of the 7,298 women who completed an oral glucose tolerance test, 54 were ineligible, 1,938 were referred for treatment and 4,348 had normal tolerance tests. Thus 958 with abnormal tolerance tests had mild GDM and were randomized.
Groups:
- Nutritional Counseling & Self Blood Glucose Monitoring: Within one week of enrollment, women in the treatment group receive formal nutritional counseling and will be instructed on the technique of self blood glucose monitoring using a memory-based reflectance meter.
  nutritional counseling
  self blood glucose monitoring
Period: Original Trial
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Started | 485 | 473
Completed | 460 | 440
Not Completed | 25 | 33
Not completed — Lost to Follow-up | 25 | 33
Period: Follow-up Study at 5-10 Years
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Started | 460 | 440
Completed | 264 | 236
Not Completed | 196 | 204
Not completed — Not eligible or did not consent | 196 | 204

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment | Total
Number analyzed (Participants) | 485 | 473 | 958
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.7) | 28.9 (5.6) | 29.1 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 485 | 473 | 958
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Groups: Black | 56 | 54 | 110
  Ethnic Groups: White | 123 | 119 | 242
  Ethnic Groups: Asian | 22 | 28 | 50
  Ethnic Groups: Hispanic | 281 | 265 | 546
  Ethnic Groups: Other | 3 | 7 | 10
Primigravida [Count of Participants; unit: Participants] | 104 | 123 | 227
Smoking [Count of Participants; unit: Participants] | 38 | 31 | 69
Alcohol Use [Count of Participants; unit: Participants] | 23 | 11 | 34
Body-mass Index at Entry [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (5.0) | 30.2 (5.1) | 30.1 (5.0)
Glucose level after 50-g glucose-loading test - mg/dL [Mean (Standard Deviation); unit: mg/dL] | 159.0 (15.3) | 159.7 (15.5) | 159.3 (15.4)
Duration of gestation randomization [Mean (Standard Deviation); unit: weeks] | 28.8 (1.6) | 28.9 (1.5) | 28.8 (1.6)
Glucose levels in 3-hr Oral Glucose Tolerance Test (OGTT) -mg/dL [Mean (Standard Deviation); unit: mg/Dl]
  Fasting | 86.6 (5.7) | 86.3 (5.7) | 86.5 (5.7)
  1-hour | 191.8 (21.9) | 193.4 (19.3) | 192.6 (20.6)
  2-hour | 173.7 (21.8) | 173.3 (19.6) | 173.5 (20.7)
  3-hour | 137.3 (29.0) | 134.1 (31.5) | 135.7 (30.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Neonatal Morbidity
Description: The composite perinatal outcome included stillbirth, neonatal death, hypoglycemia, hyperbilirubinemia, elevated cordblood C-peptide level, and birth trauma.
Time Frame: Delivery through discharge of infant from hospital up to 120 days
Population: The results of some blood tests were not available either because samples were not obtained or were not obtained according to protocol or because they could not be assayed owing to a laboratory processing error. Data were not available in some cases because some women delivered at outside institutions.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 485 | 473
Participants
  Composite End Point Total: number analyzed (Participants) | 460 | 440
  Composite End Point Total | 149 | 163
  Hypoglycemia: number analyzed (Participants) | 381 | 357
  Hypoglycemia | 62 | 55
  Hyperbilirubinemia: number analyzed (Participants) | 450 | 418
  Hyperbilirubinemia | 43 | 54
  Elevated cord-blood C-peptide level: number analyzed (Participants) | 423 | 403
  Elevated cord-blood C-peptide level | 75 | 92
  Stillbirth or Neonatal Death | 0 | 0
  Birth Trauma: number analyzed (Participants) | 476 | 455
  Birth Trauma | 3 | 6
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; For Total Composite End Point; Test type: Superiority or Other; p = 0.14, Chi-squared; Risk Ratio (RR) = 0.87, 97% CI 2-sided [0.72 to 1.07]
Statistical Analysis 2: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Analysis for Hypoglycemia; Test type: Superiority or Other; p = 0.75, Chi-squared; Risk Ratio (RR) = 1.06, 97% CI 2-sided [0.73 to 1.53]
Statistical Analysis 3: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Analysis for hyperbilirubinemia; Test type: Superiority or Other; p = 0.12, Chi-squared; Risk Ratio (RR) = 0.74, 97% CI 2-sided [0.49 to 1.12]
Statistical Analysis 4: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Analysis for elevated cord-blood C-peptide level; Test type: Superiority or Other; p = 0.07, Chi-squared; Risk Ratio (RR) = 0.78, 97% CI 2-sided [0.57 to 1.05]
Statistical Analysis 5: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Analysis for birth trauma; Test type: Superiority or Other; p = 0.33, Chi-squared; Risk Ratio (RR) = 0.48, 97% CI 2-sided [0.10 to 2.20]

2. Primary Outcome: Number of Children at the 5-10 Year Followup With BMI ≥ 95th Percentile for Age and Sex
Description: Number of children with BMI ≥ 95th percentile for age and sex. BMI is measured as kg / m^2. Standards based on the 2000 Centers for Disease Control growth charts.
Time Frame: Age 5-10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 264 | 236
Participants | 55 | 54
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.68 to 1.28]

3. Secondary Outcome: Number of Neonates Who Were Large for Gestational Age at Delivery
Time Frame: From time of randomization through delivery (up to 17 weeks)
Population: There were 8 women in the treatment group and 19 women in the control group for whom at least some delivery data were missing
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 477 | 454
Participants | 34 | 66
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 0.49, 97% CI 2-sided [0.32 to 0.76]

4. Secondary Outcome: Number of Neonates With Macrosomia (Birth Weight > 4000 gm)
Time Frame: Assessed at Delivery
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 477 | 454
Participants | 28 | 65
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 0.41, 97% CI 2-sided [0.26 to 0.66]

5. Secondary Outcome: Number Participants Who Delivered Preterm
Description: Number of preterm deliveries before 37 weeks gestation
Time Frame: Delivery before 37 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 477 | 455
Participants | 45 | 53
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.27, Chi-squared; Risk Ratio (RR) = 0.81, 97% CI 2-sided [0.53 to 1.23]

6. Secondary Outcome: Mean Neonatal Fat Mass at Delivery
Time Frame: Assessed at delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 485 | 473
grams | 427.0 (197.9) | 464.3 (222.3)
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Neonates Who Were Small for Gestational Age
Description: Birth weight below the 10th percentile
Time Frame: From time of randomization through delivery (up to 17 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 477 | 455
Participants | 36 | 29
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.49, Chi-squared; Risk Ratio (RR) = 1.18, 97% CI 2-sided [0.70 to 1.99]

8. Secondary Outcome: Mean Neonatal Birth Weight
Description: Birth weight in grams
Time Frame: Assessed at delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 485 | 473
grams | 3302 (502.4) | 3408 (589.4)
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Infants Admitted to NICU
Description: Admission to the Neonatal Intensive Care Unit
Time Frame: Delivery through hospital discharge up to 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 477 | 455
Participants | 43 | 53
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.19, Chi-squared; Risk Ratio (RR) = 0.77, 97% CI 2-sided [0.51 to 1.18]

10. Secondary Outcome: Number of Neonates Who Received Intravenous Glucose Treatment
Description: Number of neonates who received intravenous glucose treatment at any time from delivery through hospital discharge.
Time Frame: Delivery through hospital discharge up to 120 days
Population: Data was missing for 10 infants in the treatment group and 18 infants in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 475 | 455
Participants | 25 | 31
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.32, Chi-squared; Risk Ratio (RR) = 0.77, 97% CI 2-sided [0.44 to 1.36]

11. Secondary Outcome: Number of Neonates Who Experienced Respiratory Distress Syndrome
Description: Number of neonates who experienced Respiratory Distress Syndrome at any time from delivery through hospital discharge
Time Frame: Delivery through hospital discharge up to 120 days
Population: Data was missing for 8 infants in the treatment group and 18 infants in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 477 | 455
Participants | 9 | 13
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.33, Chi-squared; Risk Ratio (RR) = 0.66, 97% CI 2-sided [0.26 to 1.67]

12. Secondary Outcome: Number of Participants Who Underwent Labor Induction
Description: Number of participants who underwent labor induction
Time Frame: From time of randomization through induction (up to 17 weeks)
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
Participants | 130 | 122
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.86, Chi-squared; Risk Ratio (RR) = 1.02, 97% CI 2-sided [0.81 to 1.29]

13. Secondary Outcome: Number of Participants Who Underwent Cesarean Delivery
Description: Delivery by cesarean section
Time Frame: Delivery
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
Participants | 128 | 154
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 0.79, 97% CI 2-sided [0.64 to 0.99]

14. Secondary Outcome: Number of Neonates Who Experienced Shoulder Dystocia
Description: Number of neonates who experienced shoulder dystocia during labor and delivery
Time Frame: During the process of labor through delivery
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
Participants | 7 | 18
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 0.37, 97% CI 2-sided [0.14 to 0.97]

15. Secondary Outcome: Number of Participants Who Experienced Preeclampsia
Description: Number of participants who experienced preeclampsia
Time Frame: From time of randomization through delivery (up to 17 weeks)
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
Participants | 12 | 25
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 0.46, 97% CI 2-sided [0.22 to 0.97]

16. Secondary Outcome: Number of Participants Who Had Preeclampsia or Gestational Hypertension
Description: Number of participants who had Preeclampsia or gestational hypertension
Time Frame: From time of randomization through delivery (up to 17 weeks)
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
Participants | 41 | 62
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.01, Chi-squared; Risk Ratio (RR) = 0.63, 97% CI 2-sided [0.42 to 0.96]

17. Secondary Outcome: Mean Maternal Body-mass Index at Delivery
Description: Mean maternal body-mass index at the time of delivery
Time Frame: Delivery
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
kg/m^2 | 31.3 (5.2) | 32.3 (5.2)
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Mean Maternal Weight Gain
Description: Mean Maternal weight gain from enrollment in the trial until delivery
Time Frame: From time of randomization through delivery (up to 17 weeks)
Population: Data was missing for 9 women in the treatment group and 18 women in the control group.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 476 | 455
kilograms | 2.8 (4.5) | 5.0 (3.3)
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Number of Children With BMI ≥ 85th Percentile for Age and Sex
Description: Number of children with BMI ≥ 85th percentile for age and sex at the 5-10 year follow-up. BMI is measured as kg/m^2. Standards base on the 2000 Centers for Disease Control growth charts.
Time Frame: Age 5-10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 264 | 236
Participants | 86 | 91
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.71 to 1.10]

20. Secondary Outcome: Number of Children at 5-10 Year Follow up With Waist Circumference >90th Percentile for Age, Sex and Race/Ethnicity
Description: Child waist circumference >90th percentile for age, sex and race/ethnicity based on a study examining cross-sectional data from the Third National Health and Nutrition Examination Survey (NHANES III)
Time Frame: Age 5-10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 264 | 236
Participants | 31 | 27
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.65 to 1.69]

21. Secondary Outcome: Number of Children at 5-10 Year Follow up With Hypertension ≥ 95th Percentile for Age, Sex and Height
Description: Hypertension ≥ 95th percentile for age, sex and height based on the National Heart, Lung and Blood Institute Expert Panel on Integrated Guidelines for Children and Adolescents.
Time Frame: Age 5 - 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 264 | 236
Participants | 30 | 23
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority; Risk Ratio (RR) = 1.23, 95% CI 2-sided [0.74 to 2.05]

22. Secondary Outcome: Number of Children at 5-10 Year Follow-up With Impaired Fasting Glucose ≥100 mg/dL
Description: Number of children at 5-10 year follow-up with impaired fasting glucose ≥100 mg/dL
Time Frame: Age 5-10 years
Population: The number of children for whom glucose data is available is 390, lower than the larger follow-up sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 210 | 180
Participants | 12 | 13
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.36 to 1.62]

23. Other Pre Specified Outcome: Mean Gestational Age at Birth
Description: Mean Gestational age at the time of delivery
Time Frame: Delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Number analyzed (Participants) | 485 | 473
weeks | 39.0 (1.8) | 38.9 (1.8)
Statistical Analysis 1: Comparison: Nutritional Counseling & Self Blood Glucose Monitoring vs No Treatment; Test type: Superiority or Other; p = 0.87, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Data on adverse events for the parent trial was collected from the time of randomization (as early as 24 weeks gestation), through delivery and up to hospital discharge of the infant, death of the infant or 120 days if still hospitalized. Data on adverse events for the follow-up study was collected at the time of the study visit when the child(ren) of the participants were 5-10 years of age.
Arm/Group | Nutritional Counseling & Self Blood Glucose Monitoring | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/485 | 0/473
Other Adverse Events (participants affected / at risk) | 0/485 | 0/473

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No